CLINICAL TRIAL: NCT00303459
Title: Effects of Combination of Bosentan and Sildenafil Versus Sildenafil Monotherapy on Morbidity and Mortality in Symptomatic Patients With Pulmonary Arterial Hypertension - A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group, Prospective, Event Driven Phase IV Study
Brief Title: Effects of the Combination of Bosentan and Sildenafil Versus Sildenafil Monotherapy on Pulmonary Arterial Hypertension (PAH)
Acronym: Compass-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-052-414; COMPASS-2 (Other: Actelion Pharmaceuticals Ltd)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: sildenafil; Combination Drug Therapy; bosentan; Pulmonary Hypertension; Pulmonary Arterial Hypertension; Multicenter Study; Antihypertensive Agents; Tracleer; endothelin receptor antagonist; Randomized Controlled Trial; Phosphodiesterase type 5 inhibitor (PDE5i); Outcome Assessment
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Bosentan
  Interventions: Drug: bosentan
- B (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bosentan — bosentan/62.5 mg tablet/b.i.d. for 4 weeks then bosentan/125 mg tablet/b.i.d.
  Arms: A
Drug: placebo — Matching bosentan placebo/b.i.d.
  Arms: B

SUMMARY:
COMPASS-2 is a Phase 4, prospective, randomized, double-blind, placebo-controlled, event-driven study evaluating the effect of bosentan on the time to first confirmed morbidity/mortality event in patients with symptomatic PAH already receiving sildenafil therapy. Patients must have been receiving doses of sildenafil equal to or greater than 20 mg t.i.d. for at least 12 weeks prior to being randomized.

The study continued until the predefined target number of morbidity/mortality events was reached.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-mandated procedure
2. Males or females >=12 years of age (except for countries where this age limit is contrary to specific regulatory requirements).

   - Women of childbearing potential must have a negative pretreatment pregnancy test and must use a reliable method of contraception during study treatment and for at least 3 months after study treatment termination.

   ·Reliable methods of contraception are:

   O Barrier type devices (e.g., female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.

   O Intrauterine devices. O Oral, transdermal, injectable or implantable contraceptives only in combination with a barrier method.
   * Hormone-based contraceptives alone, regardless of the route of administration, are not considered as reliable methods of contraception.
   * Abstention, rhythm method, and contraception by the partner alone are not acceptable methods of contraception.

     * Women not of childbearing potential are defined as postmenopausal (i.e., amenorrhea for at least 1 year), or documented surgically or naturally sterile.
3. Patients with symptomatic PAH
4. Patients with the following types of PAH belonging to WHO Group I:

   * Idiopathic (IPAH)
   * Familial (FPAH)
   * Associated with (APAH):

     i. Collagen vascular disease with normal left ventricular function (ejection fraction (EF) > 50%) ii. Congenital systemic-to-pulmonary shunts at least 2 years post surgical repair iii. Drugs and toxins
5. PAH diagnosed by right heart catheter showing:

   * Mean pulmonary arterial pressure (mPAP) >= 25 mm Hg AND
   * Pulmonary capillary wedge pressure (PCWP) =< 15 mm Hg or left ventricular end diastolic pressure (LVEDP) =< 15 mmHg If both PCWP and LVEDP are available then the LVEDP value is retained for inclusion.
6. Treatment with a stable dose of sildenafil equal to or greater than 20 mg t.i.d. for at least 12 weeks prior to randomization (no sildenafil dosage adjustment should occur in this period) 7)150 m =< 6-minute walk test (6MWT) =< 480 m, documented by 2 tests with second 6MWT within 15% of first 6MWT distance or a third test required

Exclusion Criteria :

1. PAH belonging to WHO group II-V
2. PAH associated with portal hypertension and HIV infection
3. PAH associated with thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders and splenectomy
4. PAH associated with significant venous or capillary involvement (PCWP > 15 mmHg): pulmonary veno-occlusive disease and pulmonary capillary hemangiomatosis
5. Persistent pulmonary hypertension of the newborn
6. Significant valvular disease with valvular lesions to be excluded by echocardiogram within 2 years prior to randomization (i.e. patients with tricuspid or pulmonary insufficiency secondary to PAH can be included)
7. Restrictive lung disease: total lung capacity (TLC) < 60% of normal predicted value (see Appendix 3)
8. Obstructive lung disease: forced expiratory volume/forced vital capacity (FEV1/FVC) < 0.5
9. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
10. Known HIV infection
11. Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements or that may interfere with the safety or the evaluation of the study, such as chronic infection, chronic renal failure etc.
12. Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
13. Pregnancy or breast-feeding
14. Condition that prevents compliance with the protocol or adherence to therapy
15. Systolic blood pressure < 85 mmHg
16. Body weight < 40 kg
17. Hemoglobin <75% of the lower limit of the normal range
18. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal ranges
19. Known hypersensitivity or history of drug-related adverse events with bosentan (e.g. increase in liver function test results), or any of the excipients of its formulation
20. Receipt of an investigational product other than sildenafil within 3 months before start of study treatment
21. Treatment with endothelin receptor antagonists (ERAs), prostanoids or phosphodiesterase (PDE) 5 inhibitors other than sildenafil within 3 months prior to randomization
22. Concomitant systemic treatment within 1 week prior to randomization with

    * calcineurin inhibitors (e.g., cyclosporine A and tacrolimus), sirolimus and everolimus
    * glibenclamide (glyburide)
    * both cytochrome P2C9 (CYP2C9) and cytochrome P3A4 (CYP3A4) (e.g., fluconazole, amiodarone, voriconazole)
    * combination of drugs that inhibit CYP2C9 and CYP3A4
23. Treatment with nitrates and alpha-blockers at time of randomization
24. In the opinion of the investigator - patients in need for treatment with any prostanoid up to Visit 4
25. Significant left ventricular dysfunction

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2006-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

REFERENCES:
- [Derived] McLaughlin V, Channick RN, Ghofrani HA, Lemarie JC, Naeije R, Packer M, Souza R, Tapson VF, Tolson J, Al Hiti H, Meyer G, Hoeper MM. Bosentan added to sildenafil therapy in patients with pulmonary arterial hypertension. Eur Respir J. 2015 Aug;46(2):405-13. doi: 10.1183/13993003.02044-2014. Epub 2015 Jun 25. PMID 26113687
- See also: Tracleer for PAH approval page at Drugs@FDA.gov — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject, first visit was17 May 2006 and last subject, last visit was 05 Dec 2013.
Pre-assignment Details: There was a screening period of up to 14 days to assess eligibility. A total of 377 patients were screened.
Groups:
- Bosentan: Bosentan
  bosentan: bosentan/62.5 mg tablet, twice a day (b.i.d.) for 4 weeks then bosentan/125 mg tablet/b.i.d.
- Placebo: Placebo
  placebo: Matching bosentan placebo/b.i.d.
Period: Overall Study
Arm/Group | Bosentan | Placebo
Started | 159 | 175 (One subject randomized to placebo did not receive study treatment)
Completed | 76 | 86
Not Completed | 83 | 89
Not completed — Death | 33 | 44
Not completed — Withdrawal of consent | 32 | 26
Not completed — Lost to Follow-up | 5 | 4
Not completed — Administrative reason | 7 | 7
Not completed — Decision by the investigator | 5 | 7
Not completed — Lung transplantation | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized set
Groups:
- Bosentan: Bosentan
  bosentan: bosentan/62.5 mg tablet/b.i.d. for 4 weeks then bosentan/125 mg tablet/b.i.d.
- Total: Total of all reporting groups
Arm/Group | Bosentan | Placebo | Total
Number analyzed (Participants) | 159 | 175 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.44) | 54.7 (15.73) | 53.9 (15.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 128 | 253
  Male | 34 | 47 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 147 | 149 | 296
  Black | 7 | 12 | 19
  Hispanic | 5 | 6 | 11
  Other | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  Brazil | 36 | 35 | 71
  Czech Republic | 12 | 15 | 27
  Denmark | 3 | 4 | 7
  Germany | 19 | 22 | 41
  Greece | 4 | 5 | 9
  Portugal | 3 | 0 | 3
  Saudi Arabia | 0 | 1 | 1
  Slovakia | 4 | 3 | 7
  Spain | 1 | 1 | 2
  Sweden | 4 | 5 | 9
  United Kingdom | 0 | 1 | 1
  United States | 73 | 83 | 156

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Morbidity/Mortality Event up to the End of Study
Description: Kaplan-Meier estimate of percentage of participants without a morbidity/mortality event. A morbidity/mortality event is defined as the occurrence of a) death, b) hospitalization for worsening or complication of PAH or intravenous prostanoid initiation, c) atrial septostomy, d) lung transplantation, or e) worsening PAH, defined as "moderately" or "markedly" worsened PAH symptoms using a patient global self-assessment (PGSA) scale AND initiation of inhaled or subcutaneous prostanoids or the disease progression package (open-label bosentan). If a patient replied "no change" or "mildly worse" on the PGSA, a decrease in 6MWT of 20% versus last visit or 30% versus baseline is also required to confirm the event.
Time Frame: From baseline to end of study, approximately 86 months
Population: All randomized set
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
percentage of participants-Kaplan Meier
  Kaplan-Meier estimate at Month 4 | 96.1 | 90.6
  Kaplan-Meier estimate at Month 8 | 90.5 | 83.0
  Kaplan-Meier estimate at Month 12 | 82.7 | 74.0
  Kaplan-Meier estimate at Month 16 | 74.7 | 71.0
  Kaplan-Meier estimate at Month 20 | 71.8 | 66.1
  Kaplan-Meier estimate at Month 24 | 66.6 | 61.5
  Kaplan-Meier estimate at Month 28 | 65.8 | 55.0
  Kaplan-Meier estimate at Month 32 | 62.4 | 52.7
  Kaplan-Meier estimate at Month 34 | 57.5 | 48.8
  Kaplan-Meier estimate at Month 40 | 56.4 | 48.0
  Kaplan-Meier estimate at Month 44 | 50.6 | 46.2
  Kaplan-Meier estimate at Month 48 | 46.7 | 45.2
  Kaplan-Meier estimate at Month 52 | 45.1 | 45.2
  Kaplan-Meier estimate at Month 56 | 45.1 | 42.6
  Kaplan-Meier estimate at Month 60 | 45.1 | 39.7
  Kaplan-Meier estimate at Month 64 | 45.1 | 39.7
  Kaplan-Meier estimate at Month 68 | 40.1 | 39.7
  Kaplan-Meier estimate at Month 72 | 40.1 | 39.7
  Kaplan-Meier estimate at Month 76 | 40.1 | 36.1
  Kaplan-Meier estimate at Month 80 | 40.1 | 36.1
  Kaplan-Meier estimate at Month 84 | 40.1 | 36.1
  Kaplan-Meier estimate at End of Study | 40.1 | 36.1
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.2508, Log Rank; Hazard Ratio (HR) = 0.831, 97.31% CI 2-sided [0.582 to 1.187]

2. Secondary Outcome: Time to First Confirmed Death, Hospitalization for Worsening or Complication of PAH or Initiation of Intravenous Prostanoids, Atrial Septostomy, or Lung Transplantation
Description: Kaplan-Meier estimate of percentage of participants without an event of death, hospitalization (for worsening or complication of PAH or initiation of intravenous prostanoids), atrial septostomy or lung transplantation. Time to first confirmed death, hospitalization (for worsening or complication of PAH or initiation of intravenous prostanoids), atrial septostomy or lung transplantation from baseline to end of study was confirmed by an independent Clinical Endpoint Committee.
Time Frame: Baseline to end of study, approximately 86 months
Population: All randomized set
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
percentage of participants-Kaplan Meier
  Kaplan-Meier estimate at Month 4 | 97.4 | 95.3
  Kaplan-Meier estimate at Month 8 | 94.6 | 91.8
  Kaplan-Meier estimate at Month 12 | 89.6 | 88.8
  Kaplan-Meier estimate at Month 16 | 85.3 | 86.9
  Kaplan-Meier estimate at Month 20 | 82.3 | 83.8
  Kaplan-Meier estimate at Month 24 | 76.9 | 79.8
  Kaplan-Meier estimate at Month 28 | 76.1 | 74.7
  Kaplan-Meier estimate at Month 32 | 75.2 | 73.1
  Kaplan-Meier estimate at Month 36 | 72.2 | 64.4
  Kaplan-Meier estimate at Month 40 | 72.2 | 61.9
  Kaplan-Meier estimate at Month 44 | 64.2 | 60.1
  Kaplan-Meier estimate at Month 48 | 60.3 | 58.1
  Kaplan-Meier estimate at Month 52 | 57.4 | 56.8
  Kaplan-Meier estimate at Month 56 | 53.8 | 52.7
  Kaplan-Meier estimate at Month 60 | 53.8 | 51.3
  Kaplan-Meier estimate at Month 64 | 53.8 | 51.3
  Kaplan-Meier estimate at Month 68 | 39.8 | 49.2
  Kaplan-Meier estimate at Month 72 | 39.8 | 49.2
  Kaplan-Meier estimate at Month 76 | 39.8 | 45.1
  Kaplan-Meier estimate at Month 80 | 39.8 | 45.1
  Kaplan-Meier estimate at Month 84 | 39.8 | 45.1
  Kaplan-Meier estimate at End of Study | 39.8 | 45.1
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.8385, Log Rank; Hazard Ratio (HR) = 0.963, 95% CI 2-sided [0.673 to 1.380]

3. Secondary Outcome: Change From Baseline to Week 16 in 6 Minute Walk Test (6MWT)
Description: The 6MWT is a non-encouraged test, which measures the distance covered over a 6 minute walk; the patient is instructed to walk as far as possible in a 30 m long flat corridor, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Areas were to be well ventilated with air temperature controlled between 20 °C and 23 °C (68 °F to 76 °F). The test was to be administered at the same time of day and by the same tester throughout the study. The tester measured the distance walked by non-encouraged patients during the timed 6 minute period.
Time Frame: From baseline to week 16
Population: All randomized set
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
m
  Baseline | 363 (78.5) | 358 (73.1)
  Week 16 | 370 (98.3) | 343 (107.3)
  Change from baseline | 7.2 (66.01) | -14.6 (80.42)
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.0106, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 21.8, 95% CI 2-sided [5.9 to 37.8]

4. Secondary Outcome: Number of Participants With Improved, No Change, or Worsened World Health Organisation Functional Class From Baseline to Week 16
Description: Class I: no limitation of usual physical activity (PA) which does not increase dyspnea, fatigue, chest pain, or presyncope. Class II: mild limitation of PA. No discomfort at rest. Normal PA increases dyspnea, fatigue, chest pain, or presyncope. Class III: marked limitation of PA. No discomfort at rest. Less than ordinary activity increases dyspnea, fatigue, chest pain, or presyncope. Class IV: unable to perform any PA and who may have signs of right ventricular failure. Dyspnea and/or fatigue may be present at rest and symptoms are increased by almost any PA.
Time Frame: From baseline to Week 16
Population: All randomized set
Measure: Number; unit: participants
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
participants
  Improved | 25 | 28
  No change | 121 | 130
  Worsened | 13 | 17
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Relative risk of improvement = 0.98, 95% CI 2-sided [0.60 to 1.61]

5. Secondary Outcome: Time to Death of All Causes From Baseline to End of Study
Description: Kaplan-Meier estimate of percentage of participants without a mortality event.Time to death due to any cause.
Time Frame: Baseline to End of Study, approximately 86 months
Population: All randomized set
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
percentage of participants-Kaplan Meier
  Kaplan-Meier estimate at Month 4 | 99.4 | 98.2
  Kaplan-Meier estimate at Month 8 | 98.7 | 95.8
  Kaplan-Meier estimate at Month 12 | 96.5 | 94.0
  Kaplan-Meier estimate at Month 16 | 92.8 | 92.8
  Kaplan-Meier estimate at Month 20 | 90.6 | 89.5
  Kaplan-Meier estimate at Month 24 | 89.1 | 88.2
  Kaplan-Meier estimate at Month 28 | 85.8 | 85.9
  Kaplan-Meier estimate at Month 32 | 85.8 | 84.3
  Kaplan-Meier estimate at Month 36 | 85.8 | 78.5
  Kaplan-Meier estimate at Month 40 | 85.8 | 76.8
  Kaplan-Meier estimate at Month 44 | 81.4 | 74.9
  Kaplan-Meier estimate at Month 48 | 77.7 | 71.8
  Kaplan-Meier estimate at Month 52 | 75.0 | 70.5
  Kaplan-Meier estimate at Month 56 | 70.1 | 66.4
  Kaplan-Meier estimate at Month 60 | 67.8 | 64.9
  Kaplan-Meier estimate at Month 64 | 67.8 | 64.9
  Kaplan-Meier estimate at Month 68 | 67.8 | 64.9
  Kaplan-Meier estimate at Month 72 | 67.8 | 64.9
  Kaplan-Meier estimate at Month 76 | 67.8 | 60.3
  Kaplan-Meier estimate at Month 80 | 58.1 | 60.3
  Kaplan-Meier estimate at Month 84 | 58.1 | 60.3
  Kaplan-Meier estimate at End of Study | 58.1 | 60.3
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.4974, Log Rank; Hazard Ratio (HR) = 0.855, 95% CI 2-sided [0.544 to 1.344]

6. Secondary Outcome: Adjusted Percentage Ratio From Baseline in N-terminal Pro-B-type Natriuretic Peptide (NT-pro-BNP)
Description: Blood sampling for the measurement of NT-pro-BNP was performed and the plasma concentrations of NT-pro-BNP were determined by a certified centralized laboratory.
Time Frame: Baseline to Month 20
Population: All randomized patients with a baseline and at least one post-baseline value. Assessments considered are those where at least 60% of the patients have a post-baseline value
Measure: Geometric Mean (95% Confidence Interval); unit: Adjusted percentage ratio from baseline
Groups:
- Bosentan: Bosentan
  bosentan: bosentan/62.5 mg tablet, b.i.d. for 4 weeks then bosentan/125 mg tablet/b.i.d.
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 109 | 117
Adjusted percentage ratio from baseline
  Month 1 to Baseline | 87.46 [77.12 to 99.18] | 110.02 [97.56 to 124.06]
  Month 4 to Baseline | 92.65 [81.20 to 105.72] | 113.20 [99.61 to 128.65]
  Month 8 to Baseline | 85.21 [72.58 to 100.05] | 122.87 [104.82 to 144.02]
  Month 12 to Baseline | 84.48 [71.48 to 99.83] | 132.11 [111.95 to 155.89]
  Month 16 to Baseline | 92.69 [75.75 to 113.42] | 129.92 [106.69 to 158.20]
  Month 20 to Baseline | 98.36 [79.46 to 121.75] | 143.17 [115.86 to 176.91]
  Treatment effect over 20 months | 92.54 [82.72 to 103.52] | 121.00 [108.42 to 135.05]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.0003, Repeated measures analysis; Percentage change over placebo = -23.52, 95% CI 2-sided [-33.69 to -11.79]

7. Secondary Outcome: Change From Baseline to Week 16 in Borg Dyspnea Index
Description: The Borg dyspnea index was evaluated immediately after the 6MWT to obtain a rating of dyspnea at the end of the exercise using a scale from 0 ('Nothing at all') to 10 ('Very, very severe - maximal').
Time Frame: Baseline to Week 16
Population: All randomized set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
units on a scale
  Baseline | 3.5 (1.99) | 3.7 (2.18)
  Week 16 | 3.4 (2.12) | 3.6 (2.24)
  Change from baseline | -0.09 (1.693) | -0.08 (2.035)
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.9566, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.42 to 0.39]

8. Secondary Outcome: Change From Baseline to Week 16 in the EuroQol 5 Dimensions (EQ-5D) Questionnaire Calculated Score
Description: The EQ-5D questionnaire is a patient-reported outcome consisting of a 5 dimensional descriptive system and a visual analog scale (VAS). The descriptive system asks respondents to describe their health status. Health is defined in 5 dimensions: (1) mobility, (2) self care, (3) usual activities, (4) pain or discomfort, and (5) anxiety or depression. Each dimension is divided into 3 levels, indicating (a) no problem, (b) some or moderate problems, or (c) extreme problems. Respondents record their problem(s) in each of the 5 dimensions. Combinations of these levels define a total of 243 health states. A health state defined by the descriptive system of EQ-5D can be described by a 5-digit number with full health is indicated by 11111 and poorest health state by 33333. The EQ-5D calculated score was derived by re-assigning local scores for answers to each question and combining these local scores into a global score with ranges from 0 (worst possible outcome) to 1 (best possible outcome).
Time Frame: From baseline to Week 16
Population: All randomized set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
units on a scale
  Baseline | 0.678 (0.2172) | 0.681 (0.2138)
  Week 16 | 0.662 (0.2807) | 0.645 (0.3062)
  Change from Baseline | -0.0161 (0.25232) | -0.0361 (0.26671)
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.5571, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.020, 95% CI 2-sided [-0.036 to 0.076]

9. Secondary Outcome: Change From Baseline to Week 16 in the EuroQol 5 Dimensions (EQ-5D) Visual Analogue Scale Score
Description: The EQ-5D questionnaire is a patient-reported outcome consisting of a 5 dimensional descriptive system and a visual analog scale (VAS) together with brief demographic questions. EQ-5D VAS asks respondents to rate their perception of their overall health on a vertical visual analogue scale with 'best imaginable health state' set at 100 and 'worst imaginable health state' set at 0.
Time Frame: Baseline to Week 16
Population: All randomized set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 159 | 175
units on a scale
  Baseline | 67 (17.4) | 64 (17.5)
  Week 16 | 69 (19.9) | 66 (19.9)
  Change from Baseline | 2.1 (18.83) | 2.0 (17.01)
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.4086, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.2, 95% CI 2-sided [-3.7 to 4.0]

10. Secondary Outcome: Patient Global Self Assessment (PGSA) Status at Week 16
Description: The PGSA is a questionnaire that allows the patient to compare his/her PAH status in response to the question "How do you feel about your PAH today compared with your last visit?" asked by the investigator. Patients use a seven-point scale to respond: markedly better, moderately better, mildly better, no change, markedly worse, moderately worse, or mildly worse.
Time Frame: Week 16
Population: All randomized set, patients who completed the assessment
Measure: Number; unit: participants
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 150 | 162
participants
  Markedly better | 24 | 13
  Moderately better | 23 | 30
  Mildly better | 32 | 36
  No change | 50 | 59
  Mildly worse | 16 | 15
  Moderately worse | 3 | 5
  Markedly worse | 2 | 4

ADVERSE EVENTS:
Time Frame: Up to End of Study and up to 1 day after discontinuation of study treatment, approximately 86 weeks
Description: All treated patients. Treatment emergent adverse events.
Arm/Group | Bosentan | Placebo
Serious Adverse Events (participants affected / at risk) | 73/159 | 102/174
Other Adverse Events (participants affected / at risk) | 135/159 | 147/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=159) | Placebo (N=174)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 25 | 28
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 6 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 8
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OBLITERATIVE BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 11 | 6
BRONCHITIS (Infections and infestations) | 6 | 3
GASTROENTERITIS (Infections and infestations) | 3 | 5
CELLULITIS (Infections and infestations) | 3 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0
DIVERTICULITIS (Infections and infestations) | 2 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 1
SEPSIS (Infections and infestations) | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0
DENGUE FEVER (Infections and infestations) | 1 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 1 | 0
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 | 0
HAEMATOMA INFECTION (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
BACTERAEMIA (Infections and infestations) | 0 | 1
BRONCHITIS VIRAL (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
GASTROENTERITIS CALICIVIRAL (Infections and infestations) | 0 | 1
H1N1 INFLUENZA (Infections and infestations) | 0 | 1
INFECTED DERMAL CYST (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
SEPSIS SYNDROME (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 1
TUBERCULOSIS (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 6 | 8
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 3
ATRIAL FLUTTER (Cardiac disorders) | 2 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 1
BRADYCARDIA (Cardiac disorders) | 2 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 2
COR PULMONALE (Cardiac disorders) | 1 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ACUTE RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
TRIFASCICULAR BLOCK (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 3
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
BRADYARRHYTHMIA (Cardiac disorders) | 0 | 1
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 3
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 5 | 7
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1
SUDDEN DEATH (General disorders) | 1 | 1
GENERALISED OEDEMA (General disorders) | 0 | 3
OEDEMA PERIPHERAL (General disorders) | 0 | 2
ADVERSE DRUG REACTION (General disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
DEATH (General disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 3 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 1
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 2
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
LACERATION (Injury, poisoning and procedural complications) | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
RENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
VASCULAR RESISTANCE PULMONARY INCREASED (Investigations) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 3 | 2
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 1 | 0
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 | 0
HYPERSPLENISM (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 3 | 6
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 3
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 2
CONVULSION (Nervous system disorders) | 0 | 2
HYPOAESTHESIA (Nervous system disorders) | 0 | 2
BRAIN STEM STROKE (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1
MYASTHENIA GRAVIS (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 0
DIURETIC THERAPY (Surgical and medical procedures) | 1 | 0
FINGER AMPUTATION (Surgical and medical procedures) | 1 | 0
INCISIONAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 2
CHEMOTHERAPY (Surgical and medical procedures) | 0 | 1
RADIOTHERAPY (Surgical and medical procedures) | 0 | 1
SKIN CYST EXCISION (Surgical and medical procedures) | 0 | 1
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 0 | 1
THYMECTOMY (Surgical and medical procedures) | 0 | 1
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INFLAMMATORY CARCINOMA OF THE BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BIPOLAR I DISORDER (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 1
OVARIAN MASS (Reproductive system and breast disorders) | 0 | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 2
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 1
BILIARY DYSKINESIA (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
COLLAGEN DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
CREST SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 4
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 1
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=159) | Placebo (N=174)
OEDEMA PERIPHERAL (General disorders) | 30 | 26
HEADACHE (Nervous system disorders) | 24 | 24
COUGH (Respiratory, thoracic and mediastinal disorders) | 22 | 21
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 21 | 29
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 19
DIARRHOEA (Gastrointestinal disorders) | 19 | 19
CHEST PAIN (General disorders) | 18 | 10
DIZZINESS (Nervous system disorders) | 17 | 17
NAUSEA (Gastrointestinal disorders) | 16 | 22
URINARY TRACT INFECTION (Infections and infestations) | 16 | 13
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 16 | 7
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 15 | 35
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 | 22
ANAEMIA (Blood and lymphatic system disorders) | 15 | 10
BRONCHITIS (Infections and infestations) | 14 | 18
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 20
FATIGUE (General disorders) | 13 | 19
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 13 | 8
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 12 | 6
NASOPHARYNGITIS (Infections and infestations) | 11 | 15
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 12
SINUSITIS (Infections and infestations) | 11 | 12
LIVER FUNCTION TEST ABNORMAL (Investigations) | 11 | 4
RASH (Skin and subcutaneous tissue disorders) | 10 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 | 15
ANXIETY (Psychiatric disorders) | 9 | 11
HEPATIC ENZYME INCREASED (Investigations) | 9 | 3
VOMITING (Gastrointestinal disorders) | 8 | 12
INSOMNIA (Psychiatric disorders) | 8 | 11
PNEUMONIA (Infections and infestations) | 8 | 8
FALL (Injury, poisoning and procedural complications) | 8 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 8 | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less